CLINICAL TRIAL: NCT01995617
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity of GEN-004, a Streptococcus Pneumoniae Protein Subunit Vaccine, in Adult Subjects
Brief Title: Safety and Immunogenicity Study of Prophylactic Streptococcus Pneumoniae Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genocea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GEN-004-001
Record Dates: First submitted 2013-11-19; First posted 2013-11-26 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Streptococcus Pneumoniae
Keywords: vaccine; Streptococcus pneumoniae; Strep pneumo
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose (Cohort 1) (Experimental)
  Interventions: Biological: Placebo; Biological: GEN-004 Low Dose; Biological: GEN-004 Low Dose + Adjuvant
- Mid Dose (Cohort 2) (Experimental)
  Interventions: Biological: Placebo; Biological: GEN-004 Mid Dose; Biological: GEN-004 Mid Dose + Adjuvant
- High Dose (Cohort 3) (Experimental)
  Interventions: Biological: Placebo; Biological: GEN-004 High Dose; Biological: GEN-004 High Dose + Adjuvant

INTERVENTIONS:
Biological: Placebo — normal saline, 0.5 mL per dose
Biological: GEN-004 Low Dose — The GEN-004 Low Dose contains 10µg of each of the three antigens.
  Arms: Low Dose (Cohort 1)
Biological: GEN-004 Low Dose + Adjuvant — The GEN-004 Low Dose contains 10µg of each of the three antigens in combination with 350µg of aluminum hydroxide adjuvant.
  Arms: Low Dose (Cohort 1)
Biological: GEN-004 Mid Dose — The GEN-004 Mid Dose contains 30µg of each of the three antigens.
  Arms: Mid Dose (Cohort 2)
Biological: GEN-004 Mid Dose + Adjuvant — The GEN-004 Mid Dose contains 30µg of each of the three antigens in combination with 350µg of aluminum hydroxide adjuvant.
  Arms: Mid Dose (Cohort 2)
Biological: GEN-004 High Dose — The GEN-004 High Dose contains 100µg of each of the three antigens.
  Arms: High Dose (Cohort 3)
Biological: GEN-004 High Dose + Adjuvant — The GEN-004 High Dose contains 100µg of each of the three antigens in combination with 350µg of aluminum hydroxide adjuvant.
  Arms: High Dose (Cohort 3)

SUMMARY:
GEN-004 is a combination of 3 conserved proteins from Streptococcus pneumoniae. This is a randomized, double-blind, placebo-controlled, dose escalation study. Eligible subjects (male and non-pregnant female) will be assigned sequentially to 1 of 3 dose cohorts and randomized in a 3:1:1 ratio to receive GEN-004 with adjuvant, GEN-004 without adjuvant, or placebo, respectively. Each subject will receive up to 3 doses at 4 week intervals.

Subjects will be followed for safety, tolerability, and immunogenicity for 12 months after their last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females, ages 18 to 55 years inclusive.
2. Willing and able to provide written informed consent.
3. Willing to perform and comply with all study procedures including attending clinic visits as scheduled.
4. Willing to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, vasectomy, barrier methods such as condoms, diaphragms, intrauterine devices, and licensed hormonal methods for 28 days before and 90 days after receiving Study Drug.

Exclusion Criteria:

1. Immunocompromised individuals, including those receiving immunosuppressive doses of corticosteroids (more than 20 mg of prednisone given daily or on alternative days for 2 weeks or more within 6 months prior to the first dose of Study Drug, any dose of corticosteroids within 30 days of the first dose of Study Drug, or high dose inhaled corticosteroids [> 960 µg/day of beclomethasone dipropionate or equivalent]) or other immunosuppressive agents.
2. Presence or history of autoimmune disease, regardless of current treatment.
3. Insulin dependent diabetes.
4. Positive serologic test for HIV-1 or hepatitis C infection; positive hepatitis B surface antigen (HBsAg).
5. Screening serum chemistry or hematology abnormality ≥ Grade 1.
6. Screening urinalysis abnormality ≥ Grade 2.
7. Positive urine drug screen or alcohol Breathalyzer test at Screening or on Study Day 1.
8. Other active, uncontrolled co-morbidities that, in the opinion of the Investigator would make the subject unsuitable for the study or unable to comply with the study requirements.

   NOTE: Subjects who are taking a medication to control an underlying co-morbidity may be enrolled if there have been no changes to their medication within 60 days prior to the first dose of Study Drug.
9. Any acute illness including, fever (>100.4 degrees F [> 38 degrees C]) within 3 days prior to the first dose of Study Drug.
10. Pregnant or nursing women.
11. Receipt of any investigational drug within 30 days prior to the first dose of Study Drug.
12. Receipt of blood products within 90 days prior to the first dose of Study Drug.
13. Donation of blood or plasma within 56 days prior to Screening.
14. Receipt of a live vaccine within 28 days prior or a subunit vaccine within 14 days prior to the first dose of Study Drug or planned vaccination within 30 days following the last dose of Study Drug.
15. Prior vaccination with pneumococcal vaccine.
16. History of hypersensitivity to any component of the vaccine or history of an allergic reaction to an immunization.
17. History of invasive pneumococcal disease (i.e., sepsis, meningitis or pneumonia with bacteremia).
18. History of drug or alcohol abuse that, in the opinion of the Investigator, would interfere with the subject's ability to comply with the study requirements.
19. Any other condition that, in the opinion of the Investigator would make the subject unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of GEN-004 when administered with and without aluminum hydroxide to adult subjects. | 12 months after third (last) dose

SECONDARY OUTCOMES:
To evaluate the immunogenicity of GEN-004, as measured by TH17 (IL-17) and IgG responses to the antigens, when administered with and without aluminum hydroxide. | 12 months after third (last) dose
To evaluate the durability of immune responses up to 12 months after the last dose. | 12 months after third (last) dose

CONTACTS AND LOCATIONS:
Overall Officials: Mark Matson, MD, Principal Investigator — Prism Research
Locations (1):
- Prism Research, Saint Paul, Minnesota, United States